CLINICAL TRIAL: NCT00946166
Title: Impact of Statins on Cytokine Expression in Pneumonia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC2009-183H
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Community Acquired Pneumonia; Cardiovascular Risk Factors
Keywords: pneumonia; statins; cytokines
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Control (Placebo Comparator): Subjects receive standard treatment for pneumonia and a simvastatin-like placebo
  Interventions: Drug: Placebo
- Simvastatin (Experimental): Subjects receive simvastatin in addition to standard pneumonia treatment
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — 40 mg daily in the evening for a maximum of 14 days
  Arms: Simvastatin
Drug: Placebo — Simvastatin-like placebo administered daily in the evening for a maximum of 14 days
  Arms: Placebo Control

SUMMARY:
The investigators are conducting a study to determine the effects of a cholesterol-lowering medication, called simvastatin on pneumonia. People in the study will be in the hospital because they have pneumonia. The people will also have a medical condition like heart disease, diabetes, stroke or high cholesterol for which cholesterol-lowering medication has been shown to prevent future disease and/or death but are not taking a cholesterol-lowering medication when they go to the hospital. Some people will get treated with antibiotics only and other people will get antibiotics and simvastatin while they are in the hospital. The study will compare the effects the combination of simvastatin and antibiotics has on people with pneumonia to treatment with antibiotics alone.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age,
* Chart documentation by a clinician of an initial working diagnosis of pneumonia within 24 hours of admission,
* Chest x-ray or other imaging evidence consistent with pneumonia within 48 hours of hospitalization, and
* One of the following severity criteria: pneumonia severity index class III or higher, at least 2/5 components of the CURB-65, or ICU level care within 24 hours of admission.
* Having one Food and Drug Agency approved indication for statin therapy

Exclusion Criteria:

* Prior Treatment with one or more doses of a statin within 30-days prior to admission or during the current hospitalization.
* Hospitalization > 24 hours at time of the diagnosis of pneumonia.
* Hospitalization > 48 hours at time of study enrollment.
* Residence in a skilled nursing facility.
* Previously diagnosed human immunodeficiency virus infection with a current CD4 count < 200 cells/mm.
* Immunosuppression
* Patient or family decision to limit medical care ("comfort measures only").
* Known allergy to statin therapy.
* Active or planned pregnancy or breastfeeding.
* Inability to take oral medications at the time of study enrollment.
* Pre-existing liver disease or AST/ALT > 10% the upper limit of normal.
* Creatinine phosphokinase (CPK or CK) > 50% above the upper limit of normal.
* Partial ileal bypass.
* Concurrent treatment with potential interacting drugs: ketoconazole, itraconazole, amiodarone, clarithromycin, erythromycin, cyclosporine, danazol, niacin, protease inhibitors, telithromycin, verapamil, gemfiborzil, ezetimibe (Zetia), nefazodone.
* Transfer from an outside hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cytokine (TNF alpha, IL-1beta, IL-6, IL-8, IL-10) levels | enrollment, 24h, 48h, 72h, hospital discharge

SECONDARY OUTCOMES:
30-day mortality | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Mortensen, MD, Principal Investigator — University of Texas Health Science Center/ South Texas Veterans Health Care System
Locations (1):
- Audie L Murphy Memorial Veterans Hospital, San Antonio, Texas, United States